CLINICAL TRIAL: NCT06572215
Title: DYNAMic Renal Assessment: NOvel Methods to Assess KIDNEY Functional Reserve
Acronym: DYNAMO
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: KCH23-128
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Participants
  Interventions: Drug: Dapagliflozin
- Patients with hyperfiltration
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — On Day 3 to 16, participants will take 10mg dapaglifozin (SGLT-2 inhibitor) orally once daily.

SUMMARY:
This is a feasibility study to assess new, more practical ways of measuring renal reserve.

DETAILED DESCRIPTION:
Quantification of glomerular filtration rate (GFR) over time is the standard assessment of kidney function. In clinical practice, the endogenous marker, 'serum creatinine' concentration, is used as a static assessment of kidney function to estimate GFR. However, serum creatinine fails to increase until at least 50% of kidney tissue is lost,[2] thus is an inadequate indicator of early CKD.

GFR like many other physiological processes is not static and augments temporarily to stimuli such as exercise and protein intake, by up to 25% from baseline in healthy individuals.[3] Similar to cardiac function stress tests which predict adverse outcomes, inability to respond to renal stressors or 'reduced renal reserve' has been demonstrated to occur prior to development of CKD (e.g. in patients with diabetes and previous acute kidney injury (AKI)) and is associated with vulnerability to future AKI, despite the presence of apparently normal kidney function measured by serum creatinine concentration.[4] Renal reserve is lost with progressive CKD,[4] and has also been demonstrated to relate to severity of histological lesions.[5]

Current measurements of renal reserve (stimulated increase in GFR due to augmented renal blood flow above basal fasting values) involve administration of a compound that is freely filtered by the glomerulus, unaffected by tubular function and is physiologically inert, with assessment before and after an oral protein load or amino acid infusion which induces arterial vasodilation, increasing renal blood flow and GFR

The study proposes a comparison of two novel methods of 'dynamic renal function testing' with renal reserve testing.

ELIGIBILITY:
Inclusion:

Patients with sickle cell nephropathy, diagnosed clinically or histologically. Sickle Cell patients will be confirmed Hb SS and eGFR (CKD-EPI) ≥ 135 ml/min/1.73m2 OR Previous living kidney donation Age ≥ 4No contraindication or known allergy to any trial medications. Willing and able to provide written informed consent

Exclusion:

Aged < 40 Unable or unwilling to provide informed consent Breastfeeding or pregnant women Patients involved in other interventional research studies.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: : 44 Participants
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in eGFR from baseline to 2hours after oral protein load | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No